CLINICAL TRIAL: NCT06350630
Title: Therapeutic Effect of Hydroxychloroquine on Immunoglobulin A (IgA)Nephropathy Course QUIgAN Study
Brief Title: Therapeutic Effect of Hydroxychloroquine on Immunoglobulin A (IgA) Nephropathy Course QUIgAN Study
Acronym: QUIgAN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20PH284; 2024-512653-25-00 (EU CTIS Number)
Record Dates: First submitted 2024-03-28; First posted 2024-04-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: IgA Nephropathy
Keywords: Hydroxychloroquine; proteinuria
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: double blind trial randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Experimental): Active hydroxychloroquine once daily by oral route at 6.5 mg/kg of ideal weight/day, with maximal dose of 400/mg day
  Interventions: Drug: Hydroxychloroquine Oral Tablet
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydroxychloroquine Oral Tablet — Active hydroxychloroquine once daily by oral route at 6.5 mg/kg of ideal weight/day, with maximal dose of 400mg/day for 3 years
  Arms: Hydroxychloroquine
Drug: Placebo oral tablet — placebo once daily by oral route (no active drug - same dosage as hydroxychloroquine )
  Arms: Placebo

SUMMARY:
immunoglobulin A (IgA) nephropathy (Berger disease) is the most frequent primary glomerulonephritis worldwide. This disease accounts for about 5% of the causes of end stage renal disease in France, representing a major public health issue. Its pathophysiology seems to be triggered by mucosal immunity abnormalities leading to the systemic misaddressing of mucosal IgA, generation of circulating immunoglobulin A1 (IgA1) immune complexes finally deposited in renal glomeruli leading to renal tissue inflammation and scarring processes. Among this pathogeny, innate immunity is involved at several steps, including mucosal immunity.

In this regard, hydroxychloroquine has been shown to generate a global anti-inflammatory effect, particularly through its action on Toll like receptors and dendritic cells. This drug is well tolerated, widely used for other auto-immune diseases (e.g. Systemic Lupus Erythematosus) and very low priced.

One randomized controlled study conducted in China has recently shown a significant drop in proteinuria of IgA nephropathy patients treated with hydroxychloroquine (-48.4%) compared to the placebo group (+10.0%), after a quite short-term follow-up (6 months) and a moderate statistical power (30 patients in each group).

Considering (i) the potential mechanism of therapeutic effect on this disease, (ii) the well documented safety profile of the drug for rheumatologic indications and posologies, and its low cost (iii) its efficacy in reducing proteinuria in IgA nephropathy patients in a preliminary Chinese randomized control study, the investigators aim in this study at establishing the beneficial impact of hydroxychloroquine on IgA nephropathy in a double blind randomized controlled trial on a Caucasian French population with harder outcomes and a longer follow-up compared to the Chinese preliminary study.

ELIGIBILITY:
Inclusion Criteria:

* Social security affiliation
* Signed informed consent
* With biopsy proven IgA nephropathy (any vintage)
* With at least one Oxford lesion (M, E, S, T, C) on last available kidney biopsy - With urine albumin/creatinine > 300mg/g,
* under maximal tolerated labeled dose of renin-angiotensin-aldosterone system (RAAS) inhibitors for at least 3 months
* Sodium-Glucose Transport Protein 2 (SGLT-2) inhibitors initiated at least 1 month before inclusion visit
* Only patients treated with SGLT2i and RAAS dual therapy before inclusion
* With estimate GFR above 15 mL/min/1,73m² (Chronic Kidney Disease - EPIdemiology collaboration CKD-EPI formula)
* Woman in childbearing with a highly effective method of contraception
* Agreement of woman in childbearing potential (WOCBP) to perform a urine pregnancy test every month until three months after the end of study treatment
* Agreement of fertile male with WOCBP partner to use a condom for the duration of the study treatment up to 3 months after treatment the end of study treatment.

Exclusion Criteria:

* Secondary IgA nephropathy (Henoch Schonlein purpura, cirrhosis, inflammatory bowel disease)
* Corticosteroid or immunosuppressive therapies in the past year before screening
* Contra-indication to hydroxychloroquine (retinopathy, maculopathy, history of intolerance to hydroxychloroquine…)
* Uncontrolled hypertension (systolic blood pression> 160 mmHg and/or diastolic blood pression >110 mmHg )
* Long QT interval and/or QT prolonging medicines
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Absolute difference in estimate Glomerular Filtration Rate (GFR) between hydroxychloroquine group and control group evolution | 3 years

SECONDARY OUTCOMES:
nephrological follow-up: proteinuria | 1 year
nephrological follow-up: albuminuria | 1 year
nephrological follow-up: GFR | 1 year
nephrological follow-up: hematuria | 1 year
nephrological follow-up: systolic and diastolic blood pressure | 1 year
nephrological follow-up: proteinuria | 2 years
nephrological follow-up: albuminuria | 2 years
nephrological follow-up: GFR | 2 years
nephrological follow-up: hematuria | 2 years
nephrological follow-up: systolic and diastolic blood pressure | 2 years
nephrological follow-up: proteinuria | 3 years
nephrological follow-up: albuminuria | 3 years
nephrological follow-up: hematuria | 3 years
nephrological follow-up: systolic and diastolic blood pressure | 3 years
end stage renal disease (GFR< 15mL/min/1.73m²) | 3 years
death | 3 years
adverse events (pruritus, gastro-intestinal disorders) and serious adverse events (QT enlargement, cardiomyopathy, ophthalmologic disorders, neuromyopathy, cytopenia) | 3 years

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU Gabriel Montpied, Clermont-Ferrand
  - Hospices Civils de Lyon, Lyon
  - AP-HM Hôpital de la Conception, Marseille
  - APHP Hôpital Bichat, Paris
  - APHP Hôpital de Tenon, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Saint-Etienne, Saint-Etienne